CLINICAL TRIAL: NCT01588847
Title: Long-term Outcome After Radical Lymph Node Dissection of Malignant Melanoma. Comparison Between Regional Versus General Anesthesia With Respect to Impact of Perioperative Immunoediting and Validation of New Potential Predictive Biomarkers
Brief Title: Anesthesia and Cancer Recurrence im Malignant Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-AnIt-11
Record Dates: First submitted 2012-03-13; First posted 2012-05-01 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Malignant Melanoma
Keywords: perioperative immunoediting; potential predictive biomarkers; lymph node dissection
MeSH Terms: conditions — Melanoma | interventions — Anesthesia, Spinal; Anesthesia, Conduction; Anesthesia, General; Sufentanil; Propofol; Rocuronium; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regional anesthesia (Experimental)
  Interventions: Procedure: Spinal anesthesia with Bupivacaine hyperbar 0.5 %
- General anesthesia (Active Comparator)
  Interventions: Procedure: General anesthesia with Sufentanil, Propofol and Rocuronium and Sevoflurane

INTERVENTIONS:
Procedure: Spinal anesthesia with Bupivacaine hyperbar 0.5 % — Spinal anesthesia with Bupivacaine hyperbar 0.5 %
  Other Names: Regional anesthesia
  Arms: Regional anesthesia
Procedure: General anesthesia with Sufentanil, Propofol and Rocuronium and Sevoflurane — General anesthesia with Sufentanil, Propofol and Rocuronium and Sevoflurane
  Other Names: General anesthesia
  Arms: General anesthesia

SUMMARY:
Studies in animals and retrospective studies in humans show that regional anesthesia reduces metastatic cancer dissemination.

The investigators hypothesize that in patients suffering from malignant melanoma who have to undergo radical inguinal lymph node dissection immune function will be less compromised and long term survival will be superior when spinal anesthesia is compared to general anesthesia.

DETAILED DESCRIPTION:
Results of basic science indicate that regional anesthesia prevents perioperative immunosuppression and reduces postoperative metastatic cancer dissemination. If this would occur in humans, optimised anesthetic management might improve long-term outcome after cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for inguinal lymph node dissection because of malignant melanoma of the lower limb
* Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Female patients who are pregnant or nursing
* Multiple organ failure
* Contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | five years

SECONDARY OUTCOMES:
Changes of the total amount of immune cells | 15 minutes before end of surgery
  Change of the total amount of T-lymphocytes, B-lymphocytes, NK-cells, activity of NK-cells, changes in TGF-beta, activation status of thrombocytes from baseline until 15 minutes before end of surgery
Changes of the total amount of immune cells | 24 hours postoperatively
  Change of the total amount of T-lymphocytes, B-lymphocytes, NK-cells, activity of NK-cells, changes in TGF-beta, activation status of thrombocytes from baseline until 15 minutes before end of surgeryfrom baseline until 24 hours postoperatively
Changes of the total amount of immune cells | Five days postoperatively
  Change of the total amount of T-lymphocytes, B-lymphocytes, NK-cells, activity of NK-cells, changes in TGF-beta, activation status of thrombocytes from baseline until 15 minutes before end of surgeryfrom baseline until 24 hours postoperatively
Potential predictive biomarkers | 15 minutes before end of surgery
  Change of potential predictive biomarkers from baseline until 15 minutes before end of surgery postoperatively
Potential predictive biomarkers | 24 hours postoperatively
  Change of potential predictive biomarkers from baseline until 24 hours postoperatively
Potential predictive biomarkers | Five days postoperatively
  Change of potential predictive biomarkers from baseline until 5 days (plus or minus 1 day) postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hugo K Van Aken, MD PhD, Study Chair — University Hospital Muenster, Department of Anesthesia, Intensive Care and Pain Therapy
Locations (1):
- Fachklinik Hornheide, Department of Anesthesiology, Intensive Care and Pain Therapy, Münster, Germany